CLINICAL TRIAL: NCT00159939
Title: Prone-Supine Study II: The Effect of Prone Positioning for Patients Affected by Acute Respiratory Distress Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Luciano Gattinoni, Policlinico Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 392
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: ARDS, Human
Keywords: ARDS; prone position
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Prone Position

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prone position (Active Comparator): prone positioning
  Interventions: Procedure: prone positioning
- supine position (No Intervention)

INTERVENTIONS:
Procedure: prone positioning — prone positioning
  Arms: prone position

SUMMARY:
The purpose of this study is to determine whether prone positioning is effective in improving survival in patients affected by acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
BACKGROUND: The beneficial effect of prone positioning on arterial oxygenation has been well demonstrated in ALI/ARDS patients. Moreover prone positioning has an impact on the distribution of the lung densities. Finally, after a period of prone position, the respiratory compliance and the arterial oxygenation markedly improve compared to the pre-pronation values. Overall, these evidences suggests that the prone positioning may affect the outcome of ARDS patients. Recently we reported the effect of prone positioning on the outcome of ARDS patients. In this study the treatment consisted of 6 hours of pronation daily for the first ten days after the onset of acute respiratory failure. Although we did not find any difference of outcome in the general population of ARDS patients (at ten days, at discharge from ICU and after 6 months), a post hoc analysis identified a reduction in mortality at the end of the 10-days treatment period in the quartile of patients affected by most severe ARDS. A critical analysis of some of the methodological weaknesses of the previous study, together with the new information emerging from other studies, led to the adoption of major changes in the overall conception as well as in the operational design of the protocol:

* a substantial prolongation of the daily exposure to the prone position (from 6 up to a minimum of 20 hours);
* the abolition of a time window for the duration of treatment, which is not stopped except in coincidence with weaning of the patient;
* a predefined scheme for applying mechanical ventilation in both groups, based on the "lung protective strategy" concept.

OBJECTIVE: To assess the effect of prone positioning on mortality in ARDS patients, stratified at randomization according to predefined criteria of severity of respiratory failure.

STUDY DESIGN: This is a randomized, controlled, multi-center study. The patients will be randomized in two groups:

* Controls will receive optimised standard intensive treatment, including protective ventilatory strategy;
* Treatment: extended (at least 20 hrs) daily prone positioning is added to control treatment.

STUDY PROCEDURES: As soon as patients are assessed in terms of inclusion and exclusion criteria, they should be notified to the coordination center to be assigned to either the control or the treatment group according to a randomization scheme which includes stratification by severity of ARDS. On the basis of the respiratory failure severity at baseline, patients will be stratified as:

* Mild ARDS: 100≤PaO2/FiO2≤200 with 5≤PEEP≤10 cmH2O.
* Severe ARDS: PaO2/FiO2<100 with 5 cmH2O ≤ PEEP.

The patients enrolled in both the randomization arms will be ventilated according to a protective strategy.

The prone positioning will be preferentially performed with the RotoProne® bed.

The patients assigned to the treatment group must be put in a prone position daily:

* for at least 20 hours (any + variation >2 hrs must be motivated in the CRF)
* for up to 28 days

Major non-compliance with the randomized treatment (prone positioning for the control, and withdrawal for the intervention group) will be motivated in the CRF, and they are expected to occur only to better protect the well-being of the patients. The originally assigned randomized strategy must be re-established as soon as possible.

The end of the study treatment period is at 28 days from the randomization, or at the extubation, whichever occurs first.

DATA COLLECTION: The data collection forms will be sent to the Coordinating Center. The data should be collected at 12 hours interval (two times daily). We will perform a "Morning" assessment and a "Evening" assessment. The assessments should be done after at least 30 minutes from any manoeuvre that could affect the measurement (i.g., patient rolling for nursing, bronchoaspiration).

* Controls group: both "morning" and "Evening" assessments will be done in supine position at 12 hours interval.
* Treatment group: the "Morning" assessment should be done in supine position and after at least 45 minutes the patient is in supine position; in the "Evening" assessment, the data has to be collected in prone position and after at least 60 minutes the patient is in that position.

SAFETY ASPECTS AND SEVERE ADVERSE EVENTS (SAE) REPORTING: GCP rules will be strictly applied, including timely reporting to the study coordination within 48 hours from their occurrence of the SAEs not included in the efficacy end-points.

Clinical investigators and nurses of each of the participating centers will be instructed to monitor specifically and to document the adverse events more likely to be associated with the study treatment.

STUDY ORGANIZATION AND MONITORING: The centers which are admitted to the study have been selected on the basis of their previous involvement in multicenter clinical trials and the clinical experience in the application of prone position. These criteria will favour both the homogeneity and/or comparability of the standard background treatment, as well as the monitoring of the quality of the data.

The overall coordination of the study is the task of an interdisciplinary group which assures:

* the initial training of the investigators
* the real-time monitoring of all data foreseen in the CRF, through a close feed-back with each center;
* availability of a permanent 24 hours phone help-line, to answer clinical and operational queries originated by the centers;
* the periodical organization (at least 2/yr) of meetings among the participating teams (investigators and nurses), to ensure an interactive discussion of emerging problems;
* the overall quality control and management of the study data-base.

STATISTICAL ASPECTS: The characteristics of the trial (relative low frequency of the clinical condition, unavoidable concentration of the proning instrument in a limited number of centers, in opportunity of an excessive prolongation of the recruitment period which could coincide with important modifications of the way the background care develops) need to be considered when defining the sample size.

The primary outcome of the study is the overall mortality at 28 days from randomisation and it is used for sample size calculations. The study is planned to detect a 15 percent of absolute decrease in 28 day mortality, at a power of 80 percent, enrolling 170 patients in each arms. The main analysis will be performed according to an intention-to-treat approach.

The primary endpoint will be monitored using the sequential procedure of Peto et al. There will one interim analysis to assess efficacy, scheduled at approximately ½ of expected number of patients to be recruited. Accordingly, the corresponding significance level for evidence of benefit to stop the trial will be α=0.01.

ADMINISTRATIVE, LEGAL, ETHICAL ISSUES: The Prone-Supine 2 study is sponsored by a collaborative group, which has been active over the last ten years in conducting clinical trials in intensive care (5, 10).The study has been planned and is managed independently, and the clinicians who take active part in the study do not receive economic incentives. The RotoProne® bed is provided to each center by the producer (KCI Medical Products, San Antonio, TX, USA), who ensures also a small financial support for the study co-ordination (50.000 USD/years).

The data which are produced belong to the study group, who ensures their publication and their availability for public authorities.

All data related to the patients included in the study are treated in strict compliance with the Italian Laws related to privacy 675/1996.

The informed consent for the patients will be administered as soon as and every time the clinical conditions of the same patients are compatible with the procedure, thus following the provisions set forth by the ICH-GCP guidelines (11), and confirmed by the most recent European Directive 2001/20/CE Decreto Legislativo 211 24/06/2003. It is worth recalling that there is no legal basis for requiring the consent to a relative of the patient.

COMMITTEES:

Steering Committee L. Gattinoni, G. Tognoni; Scientific and Organizing Secretariat R. Fumagalli, R. Latini, A. Pesenti, P.Taccone; Nursing Coordination G. Saia, W. Rositani, V. Del Bello.; Data and Safety Monitoring Board R. Malacrida, M.G. Valsecchi, P. Suter; Data Management and Analysis E. Nicolis, S. Barlera;

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving mechanical ventilation will be enrolled if they meet criteria for acute respiratory distress syndrome, with the PaO2/FiO2 ratio criterion modified as follows:

  * PaO2/FiO2 ratio ≤ 200 with 5 ≤ PEEP ≤ 10 cmH2O

Exclusion Criteria:

* Age < 16 years.
* > 72 hours since all inclusion criteria are met.
* Lung transplant, liver transplant or bone marrow transplant.
* Clinical or instrumental evidence of cerebral edema or elevated endocranial pressure.
* Conditions which are thought to contraindicate the use of prone positioning (i.e., not-stabilized bone fracture, column fracture, pelvis fracture, multiple rib fracture with chest-wall instability, severe haemodynamic instability).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2004-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mortality | at 28 days

SECONDARY OUTCOMES:
Ventilator-free days | ICU discharge
Number of days without respiratory failure | ICU discharge
Number of days of dysfunction for each organ system and cumulative dysfunction (sequential organ failure assessment [SOFA] score) | ICU discharge
Mortality | at ICU discharge, at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Gattinoni, MD, FRCP, Study Director — Policlinico Hospital of Milan
Locations (17):
- Italy (17):
  - Hospital "Ospedali Riuniti di Bergamo", Bergamo
  - Hospital "Ospedale Maggiore di Bologna", Bologna
  - Hospital "di Circolo", Busto Arsizio
  - Hospital "A.Uboldo", Cernusco sul Naviglio
  - Hospital "di Circolo", Desio
  - Hospital "S.Martino", Genova
  - Hospital "Civile di Legnano", Legnano
  - Hospital "S.Paolo", Milan
  - Hospital "Sacco", Milan
  - Humanitas, Milan
  - Policlinico Hospital, Milan
  - Hospital "S.Gerardo", Monza
  - Hospital of Padova, Padua
  - Policlinico "S.Matteo", Pavia
  - Hospital "Caravaggio", Treviglio
  - Hospital "S.Bortolo", Vicenza
  - Hospital "Ospedale Civile", Vimercate

REFERENCES:
- [Background] Gattinoni L, Pelosi P, Vitale G, Pesenti A, D'Andrea L, Mascheroni D. Body position changes redistribute lung computed-tomographic density in patients with acute respiratory failure. Anesthesiology. 1991 Jan;74(1):15-23. doi: 10.1097/00000542-199101000-00004. PMID 1986640
- [Background] Pelosi P, Tubiolo D, Mascheroni D, Vicardi P, Crotti S, Valenza F, Gattinoni L. Effects of the prone position on respiratory mechanics and gas exchange during acute lung injury. Am J Respir Crit Care Med. 1998 Feb;157(2):387-93. doi: 10.1164/ajrccm.157.2.97-04023. PMID 9476848
- [Background] Langer M, Mascheroni D, Marcolin R, Gattinoni L. The prone position in ARDS patients. A clinical study. Chest. 1988 Jul;94(1):103-7. doi: 10.1378/chest.94.1.103. PMID 3383620
- [Background] Gattinoni L, Tognoni G, Pesenti A, Taccone P, Mascheroni D, Labarta V, Malacrida R, Di Giulio P, Fumagalli R, Pelosi P, Brazzi L, Latini R; Prone-Supine Study Group. Effect of prone positioning on the survival of patients with acute respiratory failure. N Engl J Med. 2001 Aug 23;345(8):568-73. doi: 10.1056/NEJMoa010043. PMID 11529210
- [Background] Bernard GR, Artigas A, Brigham KL, Carlet J, Falke K, Hudson L, Lamy M, Legall JR, Morris A, Spragg R. The American-European Consensus Conference on ARDS. Definitions, mechanisms, relevant outcomes, and clinical trial coordination. Am J Respir Crit Care Med. 1994 Mar;149(3 Pt 1):818-24. doi: 10.1164/ajrccm.149.3.7509706.
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Geller NL, Pocock SJ. Interim analyses in randomized clinical trials: ramifications and guidelines for practitioners. Biometrics. 1987 Mar;43(1):213-23. PMID 3567306
- [Background] Gattinoni L, Brazzi L, Pelosi P, Latini R, Tognoni G, Pesenti A, Fumagalli R. A trial of goal-oriented hemodynamic therapy in critically ill patients. SvO2 Collaborative Group. N Engl J Med. 1995 Oct 19;333(16):1025-32. doi: 10.1056/NEJM199510193331601. PMID 7675044
- [Background] Gattinoni L, Pelosi P, Valenza F, Mascheroni D. Patient positioning in acute respiratory failure. Chapter 47 in: Principles and practice of mechanical ventilation. Ed.: Tobin MJ, Illinois, USA.
- [Background] Mancebo J, Rialp G, Fernandez R, Gordo F, Albert RK. Prone vs supine position in ARDS patients. Results of a randomized multicenter trial. Am J Respir Crit Care Med 2003; 167: A180.
- [Background] Guidelines for Good Clinical Practice, par. 4.8. ICH Steering Committee meeting. 1 May 1996.
- [Derived] Taccone P, Pesenti A, Latini R, Polli F, Vagginelli F, Mietto C, Caspani L, Raimondi F, Bordone G, Iapichino G, Mancebo J, Guerin C, Ayzac L, Blanch L, Fumagalli R, Tognoni G, Gattinoni L; Prone-Supine II Study Group. Prone positioning in patients with moderate and severe acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2009 Nov 11;302(18):1977-84. doi: 10.1001/jama.2009.1614. PMID 19903918